CLINICAL TRIAL: NCT06088615
Title: Feasibility of Non-invasive Glucose Monitoring by Using Photothermal Deflectometry
Status: Completed | Type: Observational
Sponsor: Diamontech AG (Industry)
Collaborators: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Responsible Party: Sponsor
Other Study IDs: IfDT-2325-DE; CIV-23-08-043757 (Other: EUDAMED)
Record Dates: First submitted 2023-09-19; First posted 2023-10-18 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus Type 2; Diabetes Mellitus Type 1; Healthy
Keywords: non-invasive glucose monitoring; photothermal deflectometry
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the feasibility of non-invasive glucose monitoring by using photothermal deflectometry in the interstitial fluid of the skin on the wrist of subjects with diabetes mellitus type 1 and 2.

DETAILED DESCRIPTION:
The investigation is designed as an open, monocentric, non-randomized, single-arm, explorative study in adult subjects without diabetes and with type 1 or 2 diabetes mellitus (any therapy form).

The clinical investigation will be performed in an outpatient setting on up to three study days with up to 36 subjects. At least 6 subjects shall be included in each of the three subgroups (type 1 diabetes, type 2 diabetes, no diabetes)

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 OR type 2 diabetes OR no diabetes
* For subjects with diabetes: glycated haemoglobin (HbA1c) <10%
* Age ≥ 18 years
* Male or female or diverse
* An understanding of and willingness to follow the protocol
* Signed informed consent

Exclusion Criteria:

* Severe hypoglycemia resulting in seizure or loss of consciousness in the 3 months prior to enrollment
* Hypoglycemia unawareness
* Have extensive skin changes/diseases at the proposed measurement site (wrist and upper arm for FreeStyle Libre 3) that could interfere with the accuracy of glucose measurements.
* Female subjects: pregnancy, lactation period, lack of a negative pregnancy test (except in case of menopause, sterilization or hysterectomy)
* Serious acute or chronic disease besides diabetes mellitus or an anamnesis which might, in the opinion of the investigator, pose a risk to the subject, e.g. seizure disorder, adrenal disorder, dialysis for renal failure, cystic fibrosis, active infection
* Severe diabetes related complications (i.e. macro angiopathy, severe micro angiopathy, severe neuro-, retino- or nephropathy) when unstable (defined by event or increasing symptoms in the last 6 months) or with insufficient therapy
* Known severe tape reactions or allergies
* Any incapacity or general condition that, in the opinion of the investigator, prevents adequate compliance with the study procedures, e.g. mental or visual incapacity, tremor, language barriers, alcohol or drug misuse
* Not able to understand, write or read German
* Dependency from the sponsor or the clinical investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 36 adults with type 1 or 2 diabetes or without diabetes
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Accuracy of non-invasive glucose measurement in comparison to invasive glucose measurement | 3-13 days per subject
  The accuracy of glucose values determined by D-Base 2.0 Prototype B in comparison with Contour Next (CNXT) values (non-invasive vs invasive glucose measurement) is determined by the following specific analysis:
  * Number and percentage of D-Base 2.0 Prototype B results within ±15 mg/dl or ±15% as well as ±20 mg/dl or ±20% and ±30 mg/dl or ±30% of mean CNXT results for mean CNXT results <100 mg/dl or ≥100 mg/dl, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Kaluza M, Janik S, Lubinski T, Saita M, Lachmann P, Canini L, Lepro V, Mantele W. Clinical validation of noninvasive blood glucose measurements by midinfrared spectroscopy. Commun Med (Lond). 2025 Nov 15;5(1):509. doi: 10.1038/s43856-025-01241-7. PMID 41258444